CLINICAL TRIAL: NCT00522457
Title: Phase II Study Of The Trifunctional Bispecific Anti-HER-2/Neu x Anti-CD3 Antibody Ertumaxomab In Patients With HER-2/Neu Overexpressing (3+ Or 2+/FISH+) Metastatic Breast Cancer Progressing After Trastuzumab Treatment
Brief Title: Phase II Study With the Trifunctional Antibody Ertumaxomab to Treat Metastatic Breast Cancer After Progression on Trastuzumab Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: change in development plan, not due to safety concerns.
Sponsor: Neovii Biotech (Industry)
Collaborators: Fresenius Biotech North America (Industry)
Responsible Party: Manager of Regulatory Affairs, Fresenius Biotech North America
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IV-ERT-BC-04
Record Dates: First submitted 2007-08-28; First posted 2007-08-29 (Estimated); Results first posted 2011-04-29 (Estimated); Last update posted 2011-04-29 (Estimated); Status verified 2011-04

CONDITIONS: Metastatic Breast Cancer; Advanced Breast Cancer
Keywords: Breast Cancer; investigational drug; drug therapy; Antineoplastic Protocols; Immunotherapy; Metastatic breast cancer; Advanced breast cancer; Stage IV breast cancer; Her-2/neu expressing breast cancer; Her-2/neu; Trastuzumab refractory
MeSH Terms: conditions — Breast Neoplasms | interventions — ertumaxomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: ertumaxomab — Ertumaxomab will be intravenously administered to see if it can increase the patient's objective response rate.

SUMMARY:
This study has the purpose to demonstrate clinical efficacy of the investigational new drug ertumaxomab in patients with human epidermal growth factor receptor-2 (HER-2/neu) overexpressing (3+ or 2+ with a positive Fluorescence In Situ Hybridization (FISH) test result) metastatic breast cancer progressing after trastuzumab treatment.

Ertumaxomab is a trifunctional bispecific antibody targeting Her-2/neu on tumor cells and CD3 on T cells. Trifunctional antibodies represent a new concept for targeted anticancer therapy. This new antibody class has the capability to redirect T cells and accessory immune effector cells (e.g. macrophages, dendritic cells [DCs] and natural killer [NK] cells) to the tumor site. According to preclinical data, trifunctional antibodies activate these immune cells, which can trigger a complex anti-tumor immune response.

DETAILED DESCRIPTION:
This study is an open-label, non-randomized, uncontrolled, two-stage phase II study evaluating the efficacy and safety of ertumaxomab. Ertumaxomab will be administered three times at 7 day intervals by constant rate 3 hour intravenous (i.v.) infusions according to the following dose schedule: 10 µg (day 0); 100 µg (day 7 ± 1 day) and 100 µg (day 14 ± 1 day) (flat doses).

ELIGIBILITY:
Key Inclusion Criteria:

* Women ≥ 18 years, Negative pregnancy test at screening and life expectancy of at least 3 months
* metastatic (stage IV) and not curable adenocarcinoma of the breast
* Measurable disease, defined as at least one lesion that is measurable in one dimension (RECIST)
* HER-2 overexpression 3+ or 2+ FISH positive
* Patients must have received one prior therapy with trastuzumab as last treatment before entry into the study. If trastuzumab was given as single agent treatment, patients must have received prior chemotherapy for metastatic disease
* Trastuzumab has been discontinued before study entry
* disease had progressed during or after trastuzumab therapy
* Eastern Cooperative Oncology Group (ECOG)performance score of ≤ 2
* Adequate hematological, liver and kidney function

Key Exclusion Criteria:

* Women who are pregnant or breast feeding
* Any history or symptoms indicative of brain or central nervous system metastases
* Prior diagnosis of any malignancy not cured by surgery alone less than 5 years before study entry (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin)
* Human anti-murine antibody positive or hypersensitivity to murine proteins and any other component of the study drug
* Known autoimmune diseases, Human immunodeficiency virus (HIV), hepatitis B or C infection as well as other acute or chronic infection or other concurrent non-malignant co-morbidities that are uncontrolled
* Any concurrent chemotherapy, hormonal therapy, immunotherapy or corticoid therapy
* Concurrent antibiotic treatment
* Any concurrent investigational treatment for metastatic disease

Cardiovascular exclusion criteria:

* Unstable or uncontrolled pectorial angina
* Myocardial infarction during the last 6 months
* Valvular heart disease that requires treatment
* Cardiomyopathy (congestive, hypertrophic or restrictive)
* Acute myocarditis
* Congestive heart failure (CHF): dyspnea, clinically or radiologically diagnosed
* Left ventricular ejection fraction (LVEF)outside institution's normal range based on echocardiography at rest
* Left ventricular diameter > 56 mm based on M-mode echocardiography at rest
* Arrhythmias that require treatment (atrioventricular block II/III degree, atrial fibrillation, ventricular tachycardia)
* Poorly or uncontrolled hypertension, asthma, seizures, allergies, pulmonary dysfunction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Schwartz, MD, Principal Investigator — Dartmouth Hitchcock Medical Center/Norris Cotton Cancer Center; Lebanon, NH
Locations (5):
- United States (3):
  - Minneapolis, Minnesota
  - Lebanon, New Hampshire
  - New York, New York
- Canada (2):
  - Ottawa, Ontario
  - Montreal, Quebec

REFERENCES:
- [Background] Kiewe P, Hasmuller S, Kahlert S, Heinrigs M, Rack B, Marme A, Korfel A, Jager M, Lindhofer H, Sommer H, Thiel E, Untch M. Phase I trial of the trifunctional anti-HER2 x anti-CD3 antibody ertumaxomab in metastatic breast cancer. Clin Cancer Res. 2006 May 15;12(10):3085-91. doi: 10.1158/1078-0432.CCR-05-2436. PMID 16707606
- [Background] Ruf P, Lindhofer H. Induction of a long-lasting antitumor immunity by a trifunctional bispecific antibody. Blood. 2001 Oct 15;98(8):2526-34. doi: 10.1182/blood.v98.8.2526. PMID 11588051
- [Background] Riesenberg R, Buchner A, Pohla H, Lindhofer H. Lysis of prostate carcinoma cells by trifunctional bispecific antibodies (alpha EpCAM x alpha CD3). J Histochem Cytochem. 2001 Jul;49(7):911-7. doi: 10.1177/002215540104900711. PMID 11410615
- [Background] Zeidler R, Mysliwietz J, Csanady M, Walz A, Ziegler I, Schmitt B, Wollenberg B, Lindhofer H. The Fc-region of a new class of intact bispecific antibody mediates activation of accessory cells and NK cells and induces direct phagocytosis of tumour cells. Br J Cancer. 2000 Jul;83(2):261-6. doi: 10.1054/bjoc.2000.1237. PMID 10901380
- [Background] Zeidler R, Reisbach G, Wollenberg B, Lang S, Chaubal S, Schmitt B, Lindhofer H. Simultaneous activation of T cells and accessory cells by a new class of intact bispecific antibody results in efficient tumor cell killing. J Immunol. 1999 Aug 1;163(3):1246-52. PMID 10415020

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open-label phase 2 study evaluating the efficacy and safety of ertumaxomab for the treatment of metastatic breast cancer tumors. Ertumaxomab will be administered 3 times at 7 day intervals by constant rate 3 hour intravenous (IV) infusions according to the following dose schedule: 10 µg (day 0); 100 µg (day 7±1)and 100 µg(day14±1)(flat doses).
Pre-assignment Details: Patients were required to complete screening procedures and up to five treatment visits.
Period: Overall Study
Arm/Group | Ertumaxomab
Started | 19
Completed | 1
Not Completed | 18
Not completed — Due to disease progression | 16
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Ertumaxomab
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 12
  Canada | 7

OUTCOME MEASURES:

1. Primary Outcome: Clinical Efficacy Measured by Objective Response Rate (Best Response During the Course of the Study)
Time Frame: patients are monitored for 6 months
Population: The study was prematurely terminated, therefore no participants were analyzed. The primary endpoint was the objective response rate (ORR) to ertumaxomab (best response during the course of the study), defined as the number of patients with CR or PR according to RECIST, relative to the total population of treated patients
Measure: Number; unit: participants
Arm/Group | Ertumaxomab
Number analyzed (Participants) | 0

2. Secondary Outcome: Duration of Response
Description: The study was prematurely terminated, therefore no participants were analyzed
Time Frame: patients are monitored for 6 months
Population: The study was prematurely terminated, therefore no participants were analyzed
Measure: Number; unit: participants
Arm/Group | Ertumaxomab
Number analyzed (Participants) | 0

3. Secondary Outcome: Clinical Benefit Rate
Description: The study was prematurely terminated, therefore no participants were analyzed
Time Frame: patients are monitored for 6 months
Population: The study was prematurely terminated, therefore no participants were analyzed
Measure: Number; unit: participants
Arm/Group | Ertumaxomab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Ertumaxomab
Serious Adverse Events (participants affected / at risk) | 11/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ertumaxomab (N=19)
pyrexia (General disorders) | 4 (4)
asthenia (General disorders) | 1 (1)
infusion related reaction (General disorders) | 1 (2)
hypotension (Vascular disorders) | 4 (6)
hemoptysis (Vascular disorders) | 1 (1)
medical observation (Investigations) | 3 (11)
abscess intestinal (Gastrointestinal disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1)
bile duct obstruction (Hepatobiliary disorders) | 1 (1)
liver abscess (Hepatobiliary disorders) | 1 (1)
clostridial infection (Infections and infestations) | 1 (1)
urinary tract infection (Infections and infestations) | 1 (1)
malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
hydronephrosis (Renal and urinary disorders) | 2 (2)
renal failure (Renal and urinary disorders) | 1 (1)
ureteric obstruction (Renal and urinary disorders) | 1 (1)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
supraventricular tachycardia (Cardiac disorders) | 1 (2)
dehydration (Metabolism and nutrition disorders) | 1 (1)
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
confusional state (Nervous system disorders) | 1 (1)
somnolence (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ertumaxomab (N=19)
chills (General disorders) | 14 (27)
pyrexia (General disorders) | 13 (28)
fatigue (General disorders) | 11 (15)
pain (General disorders) | 3 (3)
chest pain (General disorders) | 2 (3)
flank pain (General disorders) | 2 (2)
flushing (General disorders) | 2 (2)
infusion related reaction (General disorders) | 2 (3)
asthenia (General disorders) | 1 (1)
lethargy (General disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 13 (21)
vomiting (Gastrointestinal disorders) | 10 (16)
abdominal pain (Gastrointestinal disorders) | 3 (5)
constipation (Gastrointestinal disorders) | 3 (3)
diarrhoea (Gastrointestinal disorders) | 3 (6)
abdominal discomfort (Gastrointestinal disorders) | 1 (1)
abdominal distension (Gastrointestinal disorders) | 1 (3)
abscess intestinal (Gastrointestinal disorders) | 1 (1)
oral pain (Gastrointestinal disorders) | 1 (1)
headaches (Nervous system disorders) | 14 (20)
dizziness (Nervous system disorders) | 2 (2)
amnesia (Nervous system disorders) | 1 (1)
confusional state (Nervous system disorders) | 1 (1)
dysgeusia (Nervous system disorders) | 1 (1)
neuropathy (Nervous system disorders) | 1 (1)
peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
photopsia (Nervous system disorders) | 1 (1)
hypotension (Vascular disorders) | 9 (16)
hpertension (Vascular disorders) | 4 (6)
hemoptysis (Vascular disorders) | 1 (1)
lymphoedema (Vascular disorders) | 1 (1)
aspartate aminotransferase increased (Investigations) | 4 (5)
alanine aminotransferase increased (Investigations) | 3 (4)
c-reactive protein increased (Investigations) | 3 (5)
medical observation (Investigations) | 3 (11)
blood alkaline phosphatase increased (Investigations) | 1 (1)
c-reactive protein (Investigations) | 1 (2)
electrocardiogram QT prolonged (Investigations) | 1 (1)
gamma-glutamyltransferase increased (Investigations) | 1 (1)
weight decreased (Investigations) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
myalgia (Musculoskeletal and connective tissue disorders) | 2 (5)
muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
anorexia (Metabolism and nutrition disorders) | 5 (7)
hypocalcaemia (Metabolism and nutrition disorders) | 2 (2)
decreased appetite (Metabolism and nutrition disorders) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 1 (1)
hypermagnesemia (Metabolism and nutrition disorders) | 1 (2)
hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
lymphopenia (Blood and lymphatic system disorders) | 4 (7)
anaemia (Blood and lymphatic system disorders) | 3 (3)
leukopenia (Blood and lymphatic system disorders) | 2 (2)
neutropenia (Blood and lymphatic system disorders) | 2 (2)
tachycardia (Cardiac disorders) | 4 (7)
sinus tachycardia (Cardiac disorders) | 2 (2)
supraventricular tachycardia (Cardiac disorders) | 1 (2)
oral herpes (Infections and infestations) | 3 (3)
clostridial infection (Infections and infestations) | 1 (1)
localised infection (Infections and infestations) | 1 (1)
upper respiratory tract infection (Infections and infestations) | 1 (1)
urinary tract infection (Infections and infestations) | 1 (1)
anxiety (Psychiatric disorders) | 2 (2)
insomnia (Psychiatric disorders) | 2 (2)
mood altered (Psychiatric disorders) | 1 (1)
somnolence (Psychiatric disorders) | 1 (1)
erythema (Skin and subcutaneous tissue disorders) | 2 (2)
hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1)
pallor (Skin and subcutaneous tissue disorders) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 1 (1)
malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3)
bile duct obstruction (Hepatobiliary disorders) | 1 (1)
jaundice (Hepatobiliary disorders) | 1 (1)
liver abscess (Hepatobiliary disorders) | 1 (1)
hydronephrosis (Renal and urinary disorders) | 2 (2)
renal failure (Renal and urinary disorders) | 1 (1)
ureteric obstruction (Renal and urinary disorders) | 1 (1)
cytokine release syndrome (Immune system disorders) | 1 (1)
oedema genital (Reproductive system and breast disorders) | 1 (1)
dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was prematurely terminated. This decision was based on strategic changes in the company's research and development program and resulted in limited patient data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Site may publish the results of the Study after such cooperative publication, or 1 year after Sponsor's final evaluation of all the Study data from all sites, whichever occurs first. Prior to any submission for publication, presentation, or communication of results or information arising from the Study, Investigator shall provide Fresenius Biotech at least 90 days for review and comment upon the manuscript or other material for such publication or presentation.